CLINICAL TRIAL: NCT00620698
Title: Electrical Impedance Myography as an Outcome Measure in ALS Clinical Trials
Brief Title: Electrical Impedance Myography as an Outcome Measure in Amyotrophic Lateral Sclerosis Clinical Trials
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Seward Rutkove, Principal Invesigator, Beth Israel Deaconess Medical Center
Other Study IDs: EIMALS
Record Dates: First submitted 2008-02-09; First posted 2008-02-21 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; motor neuron disease; outcome measure; biomarker; impedance
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS patients: Patients with clinically established amyotrophic lateral sclerosis

SUMMARY:
Trials evaluating new therapies for stopping or slowing the progression of ALS depend critically upon the use of outcome measures to assess whether a potential treatment is effective. The more effective an outcome measure, the fewer patients need to be enrolled and the shorter the trial. Many outcome measures have been used over the years, including strength assessments, breathing tests, functional status surveys, and nerve testing, but all are far from ideal. A new method, called electrical impedance myography (EIM) appears to be especially promising in that it provides very consistent data from one testing session to the next, is sensitive to the muscle deterioration that occurs in ALS, and is entirely painless and non-invasive. In this study, investigators from multiple institutions plan to compare several different outcome measures, including EIM, in approximately 120 ALS patients, with each patient being followed for a period of one year. All of these measures will be compared to one another and an assessment of their ability to detect disease progression made. Our goal will be to determine whether EIM can serve as a valuable new outcome measure, ultimately leading to substantially faster, more effective ALS trials requiring fewer patients.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probably ALS by El Escorial criteria
* Muscle strength of at 3.5 in one limb

Exclusion Criteria:

* Forced vital capacity of less than 70%
* Atypical forms of motor neuron disease (monomelic amyotrophy, primary lateral sclerosis)
* Pacemaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with amyotrophic lateral sclerosis (ALS)
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seward B Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Jeremy M Shefner, MD, PhD, Principal Investigator — Upstate Medical Center
Locations (8):
- United States (8):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Upstate Medical Center, Syracuse, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Virginia Medical Center, Charlottesville, Virginia

REFERENCES:
- [Background] Rutkove SB, Zhang H, Schoenfeld DA, Raynor EM, Shefner JM, Cudkowicz ME, Chin AB, Aaron R, Shiffman CA. Electrical impedance myography to assess outcome in amyotrophic lateral sclerosis clinical trials. Clin Neurophysiol. 2007 Nov;118(11):2413-8. doi: 10.1016/j.clinph.2007.08.004. Epub 2007 Sep 25. PMID 17897874

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ALS Patients
Started | 89
Completed | 60
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | ALS Patients
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Electrical Impedance Myography
Description: The main outcome measure was the coefficient of variation (CoV) in the rate of the decline for each measure over time. The CoV was calculated by dividing the standard deviation in the rate of decline across the group of subjects and dividing that by the mean rate of decline for the cohort. This approach was taken for each of the measures being evaluated (ALS Functional Rating Scale-Revised, Handheld dynamometry, Electrical impedance myography). The lower the CoV in the rate of decline, the more sensitive it is to identifying a potential treatment effect, since it suggests gives a measure of homogeneity of the rate of decline across the population as well as the overall rate of decline. The smaller the standard deviation across the group and the larger the mean rate of decline across the group, the lower the CoV and the fewer number of subjects needed for a potential clinical trial using that outcome measure.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Coefficient of Variation
Arm/Group | ALS Patients
Number analyzed (Participants) | 60
Coefficient of Variation | 0.55 [0.41 to 0.69]

2. Secondary Outcome: ALS Functional Rating Scale
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Coefficient of variation
Arm/Group | ALS Patients
Number analyzed (Participants) | 60
Coefficient of variation | 0.84 [0.58 to 1.1]

3. Secondary Outcome: Handheld Dynamometry
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Coefficient of variation
Arm/Group | ALS Patients
Number analyzed (Participants) | 60
Coefficient of variation | 0.925 [0.626 to 1.23]

ADVERSE EVENTS:
Arm/Group | ALS Patients
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No